CLINICAL TRIAL: NCT03919227
Title: Measurement of Resistance During UAS Insertion Procedure in RIRS: the Effects of Bladder Filling Degree and the Assessment of Ureter Injury.
Brief Title: Measurement of Resistance During UAS Insertion Procedure in RIRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guohua Zeng (Other)
Responsible Party: Sponsor-Investigator, Guohua Zeng, Vice president, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRER(78)2018
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Urolithiasis
Keywords: RIRS; Upper urinary calculi; Ureteral access sheath; Bladder filling degree; Ureteral injury
MeSH Terms: conditions — Urolithiasis; Urinary Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: empty bladder (Experimental): In group 1, investigator empty the bladder of urine with a catheter before inserting UAS.
  Interventions: Procedure: empty bladder before inserting UAS
- Group 2: natural state of bladder (Active Comparator): In group 2, investigator does not interfere with the filling degree of bladder before inserting UAS.
  Interventions: Procedure: do not interfere with the filling degree of bladder

INTERVENTIONS:
Procedure: empty bladder before inserting UAS — In group 1, investigator empty the bladder of urine with a catheter before inserting UAS, so that we can see if the empty bladder is easier for inserting UAS.
  Arms: Group 1: empty bladder
Procedure: do not interfere with the filling degree of bladder — In group 2, investigator does not interfere with the filling degree of bladder before inserting UAS, so that we can see if the filling degree of bladder has impact on the insertion of UAS.
  Arms: Group 2: natural state of bladder

SUMMARY:
Retrograde intrarenal surgery (RIRS) has been considered as the first-line choice for the management of <20mm kidney stones. Insertion of a ureteral access sheath (UAS) before RIRS surgery is currently accepted as an effective method to improve the effectiveness of surgery, but can be accompanied by serious complications. In long-term clinical practice, the investigators has found that different Bladder Filling Degree was accompanied by different Resistance During UAS Insertion Procedure in RIRS, which leads to the difference in success rate of UAS insertion.The investigator aims to perform a prospective and randomized controlled trial comparing the success rate of UAS insertion procedure under different bladder filling degree,and discuss the relationship between insertion resistance and ureter injury.

DETAILED DESCRIPTION:
Upper urinary calculi is a common disease that endangers human health, Retrograde intrarenal surgery (RIRS) has been considered as the first-line choice for the management of <20mm kidney stones. Insertion of a ureteral access sheath (UAS) before RIRS surgery is currently accepted as an effective method to improve the effectiveness of surgery, for UAS can drain irrigation to reduce renal pelvic pressure and maintain vision clear. But incorrect way to insert UAS can be accompanied by serious complications. For instance, If the ureter was not dilated by DJ stent before RIRS surgery, or ureter was relatively narrow, the insertion of UAS would encounter great resistance. Sometimes the ureter was violently pushed into UAS, it might cause ureteral perforation or avulsion. As for how to insert UAS correctly, there is no unified international standard at present. Different surgeons have different experience. In long-term clinical practice, the investigators has found that different Bladder Filling Degree was accompanied by different Resistance During UAS Insertion Procedure in RIRS, which leads to the difference in success rate of UAS insertion. In addition, there seems to be some relationship between the resistance of UAS insertion and the ureter injury in surgery. Therefore, the investigator aims to perform a prospective and randomized controlled trial comparing the success rate of UAS insertion procedure under different bladder filling degree, and discuss the relationship between insertion resistance and ureter injury.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be a suitable operative candidate for RIRS
2. Age 18 to 70 years
3. Normal renal function 4 .ASA score Ⅰ and Ⅱ

5. Single renal or ureteral stone ≤20mm or multiple stones the conglomerate diameter (additive maximal diameter of all stones on axial imaging of computed tomography) up to 20 mm

Exclusion Criteria:

1. Uncorrected coagulopathy and active urinary tract infection (UTI)
2. Severe cardiopulmonary dysfunction, can not tolerate sugery
3. Patients who underwent transplant or urinary diversion
4. Definite diagnosis of ureteral stricture or a history of stricture
5. The bladder volume is less than 100ml

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-09-12 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
UAS insertion success rate | intraoperatively
  Primary insertion of a UAS is not always successful. The ideal position of the UAS is with its distal extremity just below the ureteric-pelvic junction (UPJ). Insertion failure is defined as UAS cross the upj or do not reach the proximal ureter or the surgeon's decision to resign UAS insertion due to high resistance to the retrograde progression of the UAS along the urinary tract.

SECONDARY OUTCOMES:
Ureteral lesion grade | intraoperatively
  Base on post-ureteroscopic lesion scale (PULS), reported by Traxer O and Thomas A in 2013. UAS related ureteral injuries were divided into 5 grades according to ureteral wall anatomy. Grade 0 means no lesion found or only mucosal petechiae. Grade 1 means ureteral mucosal erosion without smooth muscle injury. Both Grade 0 and Grade 1 are considered as low-level injuries. Grade 2 means ureteral wall injury, including mucosa and smooth muscle, with adventitial preservation (periureteral fat not seen). Grade 3 means ureteral injury indicated ureteral perforation involving the full thickness of the ureteral wall, including the adventitia. Grade 4 means injury corresponded to total ureteral avulsion with complete rupture of ureteral continuity. Grade 2, 3 and 4 are high-level injuries.
resistance of UAS insertion | intraoperatively
  The dynamometer was used to measure the resistance of UAS insertion procedure in both two groups, so as to analysis the relationship between bladder filling degree and inserting resistance.
Complication rate | 1 month after removing the pigtail stent
  Complication is defined as any adverse event occurred intraoperatively or ≤1 month postoperatively, including intraoperative bleeding, postoperative pain and so on.The investigator will invaluate perioperative complications by modified Clavien system

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, Ph.D and M.D, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Department of Urology, Minimally Invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China